CLINICAL TRIAL: NCT06748157
Title: Non-Invasive Median Nerve Stimulation to Attenuate Atrial Tachyarrhythmias After Catheter Ablation for Atrial Fibrillation
Acronym: NEUROPULSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Ziv HealthCare Ltd. (Industry)
Responsible Party: Principal Investigator, Vivek Reddy, Director EP Service, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY-24-00641
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
Keywords: AFib; Neuromodulation; Prevent AFib
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant, Investigator
Masking Description: Patient and investigator are blinded, as is the statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Participants with CardiaCare RR2 (Active Comparator): Participants undergoing Neuromodulation Sessions (mNVS) and Active Median/Vagal Stimulation. Patients will receive training on the RR2 for home-care use, by study personnel either in person or via a video conference meeting. An instructional video will also be available for users.
  Interventions: Device: CardiaCare RR2
- Participants with Sham Device (Sham Comparator): Sham device will be dispensed, which will create a sensation but not provide therapy
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: CardiaCare RR2 — CardiaCare has developed a wrist band that delivers non-invasive neuromodulation to the median nerve to elicit a vagal response (Median-Vagus nerve stimulation-mVNS). The device is in the post-prototype development stage and is ready for human clinical trials. The CardiaCare RR2 device has already been approved by the IRB of the Chaim Sheba Medical Center, IL and the IL MOH (Ministry of Health) in an already completed pilot clinical trial for modulating AF.
  Arms: Participants with CardiaCare RR2
Device: Sham Device — Sham device will be dispensed, which will create a sensation but not provide therapy
  Arms: Participants with Sham Device

SUMMARY:
Determine the role of vagal/median nerve stimulation using the CardiaCare RR2 home care wearable neuromodulation system on suppressing atrial arrhythmias and related symptoms in patients who have undergone AF ablation. The study population will be comprised of adults (age ≥18 yrs.) who have undergone AF ablation for paroxysmal or persistent AF.

The study will assess the ability of neuromodulation, using the CardiaCare RR2 home care wearable, to suppress the following:

1. early (0-2 months) post-ablation arrhythmias that occur in the immediate post-ablation time period
2. AF/AT/AFL recurrences between months 2-6 post-ablation.This is a prospective, controlled, double-blind, randomized trial. The first 15 patients will not be randomized and will receive the active median/vagal stimulation only (open label).

The Study will be conducted in up to 1 clinical site in the United States. This study will have 1:1 randomization (active median/vagal stimulation vs sham). The study has been given NSR designation from FDA--NO IDE.

DETAILED DESCRIPTION:
Study will include continuous ECG assessment at 2 (0 for the first 15 patients, open label), 6 and 22 weeks from enrollment for 2 weeks (for 4 weeks at the first measurement for the first 15 patients, open label) and at least daily single lead ECG assessments throughout the follow up period. The ECG's generated can be viewed by physicians only to assess the frequency of RR2 treatments and will not be used to alter any other aspects of standard of care, including medical management, which will continue according to standard of care throughout the study. Patients and investigators will be blinded during the trial. Patients with paroxysmal or persistent AF undergoing AF ablation will be recruited post ablation procedure during hospitalization. During screening/baseline visit, eligible patients will be randomized to either an active treatment or a sham group (1:1 accordingly). The first 15 eligible patients will not be randomized and will receive the active median/vagal stimulation only (open label).

Patients will receive training on the RR2 for home-care use, by study personnel either in person or via a video conference meeting. An instructional video will also be available for users. Patients will be ordered to measure at home, 2 min ECG measurements with the RR2 system, two times a day throughout the study and when feeling symptoms suspected related to AF (AF/AT/PAC).

In addition, Patients will be instructed to perform Neuromodulation sessions with the RR2 home care device. Once a day for the first 2 weeks followed by three times per week for the remaining duration of the study. Additional treatments, up to once daily, will be added during this period in case the patient feels symptom, verified on single lead ECG and site staff.

Treatments will be conducted for a period of 6 months. During the study, the patients will continue to take Standard of care medication. Medications will be recorded throughout the study.

Patient Diary will be dispensed and or APP diary questioners will be used by the subject in order to document symptoms suspected as related to arrhythmia events.

ELIGIBILITY:
Inclusion Criteria

* Men and women ages ≥18 years
* Patients planned to undergo or undergoing AF ablation for paroxysmal or persistent AF and able to be randomized within 48 hours of the ablation procedure.
* Ability and willingness to sign an informed consent form.
* Ability and willingness to use CardiaCare RR2 device, continuous ECG monitoring, and has an available SmartPhone.

Exclusion Criteria

* Rheumatic heart disease
* Extensive atrial disease (* some patients may be determined to be screen failures following the ablation procedure).
* Moderate to severe mitral stenosis or history of mitral valve replacement
* Pacemaker or CRTD or any implanted electrical stimulating device
* Unilateral or bilateral vagotomy
* Peripheral neuropathy affecting the tested upper extremity.
* Severe heart failure (New York Heart Association Class III or IV) within 90 days.
* Recent (within 90 days) stroke or transient ischemic attack.
* Recent (within 90 days) myocardial infarction.
* Pregnancy or breast feeding.
* Life expectancy <1 year for any medical condition
* Currently enrolled in another study that would interfere with this study
* Unsuitable for participating in the study according to attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
AF/AFL occurrence | at 2-months and 6-months post-ablation procedure
  Burden of AF/AFL (defines as 30 seconds or longer) during the 2-months and 6-months period after ablation measured using ECG-patch monitoring and daily RR2 single lead ECG.

SECONDARY OUTCOMES:
Time to first Atrial tachycardia (AT) or Atrial Fibrillation (AF) recurrence | 2-month and 6-month post-ablation procedure
  Time to first AT or AF recurrence measured by CardiaCare RR2
Number of arrythmia occurrences | 2-month and 6-month post-ablation procedure
  Burden of all arrythmias between 2- and 6-months period after ablation will be measured using 2 weeks ECG-patch monitoring and daily RR2 single lead ECG.
Number of Atrial Arrythmia Symptoms | 6-month post-ablation procedure
  Difference in Atrial Arrythmia Symptoms during the 6 months period after ablation.
Time to first Atrial tachycardia (AT) or Atrial Fibrillation (AF) recurrence | 6 months post-ablation
  Time to first Atrial tachycardia (AT) or Atrial Fibrillation (AF) recurrence during the 6-months period after ablation.
Quality of Life measured using The European Heart Rhythm Association (EHRA) score | Baseline, 2-months, and 6-months
  The investigators will assess the change in EHRA symptom scale. The EHRA score ranges from 1 to 4. Higher scores indicate more severe symptoms.
Quality of Life measured using Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) Score | Baseline, 2-months, and 6-months
  The AFEQT is a questionnaire assessing quality of life and symptoms in atrial fibrillation patients. It covers four subscales: patient symptoms, daily activities, treatment concerns, and treatment satisfaction. Subscales from 0-100, with Full Scale range from 0 to 100, with higher scores indicating better quality of life and fewer symptom burdens.
Change in PAC/AT/AFL before and after treatment with RR2 | Baseline and 6-month post-ablation
  Change, such as increase or decrease, in incidence/frequency of atrial arrhythmias before and after treatment with study device.
Change in Heart Rate Variability (HRV) | Baseline and 6-month post-ablation
  Heart rate variability (HRV) is the variation in the time interval between consecutive heartbeats. Higher HRV indicates better cardiovascular function and stress resilience.
Number of ER Visits | 6-month post-ablation
Number of Hospitalizations | 6-month post-ablation
Number of Cardioversions | 6-month post-ablation
Number of Ablation Re-Do's | 6-month post-ablation

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Mohit Turagam, MD, Principal Investigator — Icahn School of Medicine at MS
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No